CLINICAL TRIAL: NCT01148576
Title: Influence of Hepatic Steatosis on the Therapeutic Effect of Entecavir in Chronic Hepatitis B Patients-A Randomized, Double-Blinded, Controlled Trial
Brief Title: Influence of Hepatic Steatosis on the Therapeutic Effect of Entecavir in Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: the first affiliated hospital, college of medicine, zhejiang university, the first affiliated hospital, college of medicine, zhejiang university
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCTZJU201001
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Hepatitis B; Hepatic Steatosis
Keywords: hepatic steatosis, chronic hepatitis B, entecavir
MeSH Terms: conditions — Hepatitis B, Chronic; Fatty Liver | interventions — entecavir; essential 303 forte; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control group (Other): patients only with chronic hepatitis B
  Interventions: Drug: entecavir
- model group (Active Comparator): patients with chronic hepatitis B and hepatic steatosis
  Interventions: Drug: entecavir
- Essentiale group (Experimental): patients with chronic hepatitis B and hepatic steatosis
  Interventions: Drug: essentiale + entecavir
- treatment group 2 (Experimental): patients with chronic hepatitis B and hepatic steatosis
  Interventions: Drug: Vitamin E + entecavir

INTERVENTIONS:
Drug: entecavir — entecavir 0.5 mg qd for 12 months
  Arms: control group
Drug: entecavir — entecavir 0.5 mg qd for 12 months
  Arms: model group
Drug: essentiale + entecavir — entecavir 0.5 mg qd for 12 months，Essentiale 2 tablets tid in the first 3 months and 1 tablets tid in the rest 9 months
  Arms: Essentiale group
Drug: Vitamin E + entecavir — entecavir 0.5 mg qd for 12 months, Vitamin E: 100 mg bid for 12 months
  Arms: treatment group 2

SUMMARY:
To investigate the influence of hepatic steatosis on the anti-viral effect of entecavir in chronic hepatitis B patients.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) affects approximately 360 million persons worldwide and is the most common cause of liver disease and affects over 10% of the general population in China. Hepatic steatosis is the main hepatic presentation of non- alcoholic fatty liver disease that is becoming another important liver disorder both in China and worldwide with economic development. It would be expected that hepatic steatosis might occur in CHB patients and recent studies show the frequency of steatosis in CHB ranges from 27% to 51%. However, the effect of steatosis on the anti-viral treatment in CHB patients is still vague. The aim of this RCT is to investigate the effect of steatosis on the therapeutic effect of entecavir in chronic hepatitis B patients. We will compare the anti-viral effect of entecavir among four groups: CHB group with entecavir therapy, CHB + steatosis group with entecavir therapy, CHB + steatosis group with entecavir + essentiale therapy and CHB + steatosis group with entecavir + vitamin E therapy. The speculated points are set as 3 months, 12 months and 15 months. Liver biopsy will be carried out at beginning and the 12th month. Other serum biochemical and viral markers are recorded as well as CT or ultrasound scan are repeated.

ELIGIBILITY:
Inclusion Criteria:

Patients should be diagnosed with chronic hepatitis B infection and hepatic steatosis

1. CHB infection

   * HBV-DNA ≥ 1×105 copies/ml；
   * HBeAg positive ；
   * ALT between the 2-10 times of the upper limit level
2. hepatic steatosis According to the "Guidelines for the assessment and management of non-alcoholic fatty liver disease in the Asia-Pacific region: executive summary", with test of CT scan or B ultrasound and confirmation of liver biopsy(in portion of patients)

Exclusion Criteria:

1. those receiving antiviral treatment before the study
2. those on hepatoxic drug treatment,
3. those consuming alcohol regularly or excessively,
4. those diagnosed of cirrhosis, anti-HCV or anti-Delta positive patients,
5. those diagnosed as having autoimmune or other metabolic liver diseases
6. those have wilson's disease, PBC, PSC, IBD and other diseases that may influence the process and effect of therapy
7. those who are pregnant, have mental disorder and were received anti-viral treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Differences in the anti-viral effect of entecavir among CHB patients and CHB + hepatic steatosis patients who received different drugs | 12 months
  The common measurement includes serum biochemistry markers (ALT, AST, GGT, CRP, PT, APTT, AMA, UA, Chol, TG, TB, DB, ALP, fasting glucose, insulin, et al), virus markers (HBs-Ag, Hbe-Ag, anti-HBc-Ab, HBV genotype, HBV- DNA copy, YMDD variation, et al), Liver CT scan or ultrasound (steatosis degree and fibrosis and changes in the histological features of liver biopsy(steatosis degree, inflammation and fibrosis).

SECONDARY OUTCOMES:
Differences in the sustained response rate to entecavir among CHB patients and CHB + hepatic steatosis patients who received different drugs and obtained anti-virus effect after 1 year treatment. | 15 months
  The common measurement includes serum biochemistry markers (ALT, AST, GGT, CRP, PT, APTT, AMA, UA, Chol, TG, TB, DB, ALP, fasting glucose, insulin, et al), virus markers (HBs-Ag, Hbe-Ag, anti-HBc-Ab, HBV genotype, HBV- DNA copy, YMDD variation, et al), Liver CT scan or ultrasound (steatosis degree and fibrosis).
Differences in the anti-viral effect of entecavir among CHB patients and CHB + hepatic steatosis patients who received different drugs in a short term. | 3 months
  The common measurement includes serum biochemistry markers (ALT, AST, GGT, CRP, PT, APTT, AMA, UA, Chol, TG, TB, DB, ALP, fasting glucose, insulin, et al), virus markers (HBs-Ag, Hbe-Ag, anti-HBc-Ab, HBV genotype, HBV- DNA copy, YMDD variation, et al), Liver CT scan or ultrasound (steatosis degree and fibrosis).

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital, college of medicine, zhejiang university, Hangzhou, Zhejaing, China